CLINICAL TRIAL: NCT04489771
Title: Phase 2 Study of MK-6482 in Participants With Advanced Renal Cell Carcinoma
Brief Title: A Study of Belzutifan (MK-6482) in Participants With Advanced Renal Cell Carcinoma (MK-6482-013)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-013; MK-6482-013 (Other: MSD); 2022-502123-21-00 (Registry Identifier: EU CT); 2020-001907-18 (EudraCT Number)
Record Dates: First submitted 2020-07-27; First posted 2020-07-28 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: Hypoxia inducible factor (HIF); Hypoxia inducible factor 1B (HIF-1B); Hypoxia inducible factor 2 alpha (HIF-2 alpha); Hypoxia inducible factor 2α (HIF-2α); Renal Cell Carcinoma (RCC); Kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan 200 mg (Experimental): Participants receive 200 mg of belzutifan by oral administration, once a day (QD), until disease progression or discontinuation.
  Interventions: Drug: Belzutifan
- Belzutifan 120 mg (Experimental): Participants receive 120 mg of belzutifan by oral administration, QD, until disease progression or discontinuation.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Oral administration
  Other Names: MK-6482; PT2977; WELIREG™

SUMMARY:
This study will compare the efficacy and safety of two doses of belzutifan in participants with advanced renal cell carcinoma (RCC) with clear cell component after prior therapy.

The primary hypothesis is that the higher dose of belzutifan is superior to the standard dose in terms of objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of locally advanced/metastatic RCC with clear cell component
* Has measurable disease per RECIST 1.1 as assessed by BICR
* Can submit an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has experienced disease progression on or after systemic treatment with an anti-programmed cell death 1 (PD-1)/Ligand 1 (L1) therapy for locally advanced or metastatic RCC. The anti-PD-1/L1 therapy may be monotherapy or in combination with other agent(s) such as anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) or vascular endothelial growth factor (VEGF) targeted- tyrosine kinase inhibitor (TKI). The immediately preceding line of treatment has to have been an anti-PD-1/L1 therapy
* Has received no more than 3 prior systemic regimens for locally advanced or metastatic RCC
* Has received only 1 prior anti-PD-1/L1 therapy for locally advanced or metastatic RCC
* Has recovered from all AEs due to previous therapies to ≤Grade 1 or baseline, with the exception of ≤Grade 2 neuropathy or endocrine-related AEs ≤Grade 2 requiring treatment or hormone replacement
* Has a Karnofsky performance status (KPS) score of at least 70% assessed within 10 days prior to the first dose of study intervention
* A male participant is eligible to participate if he is abstinent from heterosexual intercourse or agrees to use contraception during the intervention period and for at least 7 days after the last dose of study intervention
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a (woman of childbearing potential) WOCBP or a WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 30 days after the last dose of study intervention
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) within 24 hours before the first dose of study intervention

Exclusion Criteria:

* Has hypoxia (a pulse oximeter reading <92% at rest), requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] that have undergone potentially curative therapy
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction ≤6 months from Day 1 of study drug administration or New York Heart Association Class III or IV congestive heart failure
* Has moderate to severe hepatic impairment (Child-Pugh B or C)
* Has received colony-stimulating factors (eg, granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin [EPO]) ≤28 days prior to the first dose of study intervention
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (eg, gastrectomy, partial bowel obstruction, malabsorption)
* Has known hypersensitivity or allergy to the active pharmaceutical ingredient or any component of the study intervention (belzutifan) formulations
* Has received prior treatment with belzutifan or another hypoxia-inducible factor (HIF)-2α inhibitor
* Has received any type of small molecule kinase inhibitor (including investigational kinase inhibitor) ≤2 weeks before randomization
* Has received any type of systemic anticancer antibody (including investigational antibody) ≤4 weeks before randomization
* Has received prior radiotherapy ≤2 weeks prior to first dose of study intervention. Participants must have recovered from all radiation-related toxicities and not require corticosteroids
* Has had major surgery ≤3 weeks prior to first dose of study intervention
* Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (eg, bosentan, efavirenz, modafinil) inducers of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Is currently participating in a study of an investigational agent or is currently using an investigational device
* Has an active infection requiring systemic therapy
* Has active tuberculosis (TB)
* Has a diagnosis of immunodeficiency
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (HBV) or known active hepatitis C (HCV) infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not the best interest of the participant to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2026-10-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (48):
- United States (18):
  - Georgetown University Medical Center ( Site 0002), Washington D.C., District of Columbia
  - Univ of Miami- Sylvester Comprehensive Cancer Center ( Site 0023), Miami, Florida
  - Norton Cancer Institute - St. Matthews ( Site 0025), Louisville, Kentucky
  - Weinberg Cancer Institute at Franklin Square ( Site 0007), Baltimore, Maryland
  - Cancer Partners of Nebraska ( Site 0003), Lincoln, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0012), Omaha, Nebraska
  - New York Oncology Hematology P.C ( Site 0028), Albany, New York
  - Roswell Park Cancer Institute ( Site 0038), Buffalo, New York
  - Fox Chase Cancer Center ( Site 0026), Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic ( Site 0031), Sioux Falls, South Dakota
  - UT West Cancer Center ( Site 0032), Germantown, Tennessee
  - Urology Associates ( Site 0015), Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas ( Site 0004), Dallas, Texas
  - Baylor Scott & White Medical Center - Temple ( Site 0013), Temple, Texas
  - Huntsman Cancer Institute ( Site 0037), Salt Lake City, Utah
  - Inova Schar Cancer Institute ( Site 0001), Fairfax, Virginia
  - Blue Ridge Cancer Care - Roanoke ( Site 0017), Roanoke, Virginia
  - Kadlec Clinic Hematology and Oncology ( Site 0008), Kennewick, Washington
- Australia (3):
  - Macquarie University ( Site 1007), Macquarie University, New South Wales
  - Eastern Health - Box Hill Hospital ( Site 1003), Box Hill, Victoria
  - Peninsula Health Frankston Hospital ( Site 1001), Frankston, Victoria
- Belgium (5):
  - GZA Sint Augustinus ( Site 2003), Wilrijk, Antwerpen
  - Grand Hopital de Charleroi ( Site 2005), Charleroi, Hainaut
  - CHU de Liege ( Site 2002), Liège, Liege
  - UZ Gent ( Site 2004), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 2001), Leuven, Vlaams-Brabant
- Greece (3):
  - General Hospital of Athens "Alexandra" ( Site 1102), Athens, Attica
  - Athens University Hospital ATTIKON ( Site 1100), Chaïdári, Attica
  - University General Hospital of Larissa ( Site 1101), Larissa, Thessaly
- Ireland (2):
  - Cork University Hospital ( Site 9053), Cork
  - Tallaght University Hospital ( Site 9051), Dublin
- Israel (4):
  - Soroka Medical Center ( Site 4004), Beersheba
  - Rambam Medical Center ( Site 4001), Haifa
  - Rabin Medical Center ( Site 4002), Petah Tikva
  - Sourasky Medical Center ( Site 4003), Tel Aviv
- Netherlands (5):
  - Maastricht Universitair Medisch Centrum - MUMC ( Site 5001), Maastricht, Limburg
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 5003), Amsterdam, North Holland
  - Isala klinieken ( Site 5002), Zwolle, Overijssel
  - Erasmus MC ( Site 5000), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht ( Site 5004), Utrecht
- Russia (4):
  - Federal state budgetary institution Russian Research Centre of radiology and nuclear medicine ( Site, Moscow, Moscow
  - City Clinical Oncology Hospital No. 1 ( Site 6004), Moscow, Moscow
  - Clinical Research Center of specialized types medical care-Oncology ( Site 6002), Saint Petersburg, Sankt-Peterburg
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 6001), Saint Petersburg, Sankt-Peterburg
- United Kingdom (4):
  - Royal Free London NHS Foundation Trust ( Site 9003), London, England
  - Imperial College Healthcare NHS Trust ( Site 9004), London, London, City of
  - Churchill Hospital ( Site 9000), Oxford, Oxfordshire
  - Nottingham University Hospitals NHS Trust. City Hospital Campus ( Site 9001), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Agarwal N, Brugarolas J, Ghatalia P, George S, Haanen JB, Gurney H, Ravilla R, Van der Veldt A, Beuselinck B, Pokataev I, Suelmann BBM, Tuthill MH, Vaena D, Zagouri F, Wu J, Perini RF, Liu Y, Merchan J, Atkins MB. Randomized phase II dose comparison LITESPARK-013 study of belzutifan in patients with advanced clear cell renal cell carcinoma. Ann Oncol. 2024 Dec;35(12):1148-1156. doi: 10.1016/j.annonc.2024.08.2338. Epub 2024 Sep 2. PMID 39233312
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26234&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Belzutifan 200 mg: Participants received 200 mg of belzutifan by oral administration, once a day (QD), until disease progression or discontinuation.
- Belzutifan 120 mg: Participants received 120 mg of belzutifan by oral administration, QD, until disease progression or discontinuation.
Period: Overall Study
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Started | 78 | 76
Completed | 0 | 0
Not Completed | 78 | 76
Not completed — Death | 27 | 25
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participants Ongoing in Study | 50 | 51

BASELINE CHARACTERISTICS:
Groups:
- Belzutifan 200 mg: Participants received 200 mg of belzutifan by oral administration, QD, until disease progression or discontinuation.
- Total: Total of all reporting groups
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (9.8) | 61.6 (9.8) | 63.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 59 | 64 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 69 | 72 | 141
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 71 | 69 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Risk Factor [Count of Participants; unit: Participants] — Participants were stratified by their IMDC Risk Factor (favorable vs. intermediate or poor).
  Participants
    Favorable | 13 | 14 | 27
    Intermediate or Poor | 65 | 62 | 127

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who had a complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experienced a CR or PR as assessed by blinded independent central review based on RECIST 1.1 was presented.
Time Frame: Up to approximately 27 months
Population: The analysis population consisted of all randomized participants based on the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Percentage of Participants | 23.1 [14.3 to 34.0] | 23.7 [14.7 to 34.8]
Statistical Analysis 1: Comparison: Belzutifan 200 mg vs Belzutifan 120 mg; Test type: Superiority — P-value, difference in percentage and associated 95% CI were calculated using Miettinen & Nurminen method stratified by IMDC risk categories (favorable vs. intermediate or poor); p = 0.5312, Miettinen & Nurminen — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = -0.5, 95% CI 2-sided [-14.0 to 12.9] — Belzutifan 200 mg minus Belzutifan 120 mg

2. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST 1.1 as Assessed by BICR
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by blinded independent central review was presented.
Time Frame: Up to approximately 27 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Months | 9.1 [5.5 to 12.0] | 7.3 [5.6 to 9.5]
Statistical Analysis 1: Comparison: Belzutifan 200 mg vs Belzutifan 120 mg; Test type: Other; p = 0.3861, Log Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; One-sided nominal p-value based on log-rank test stratified by IMDC risk group (favorable vs. intermediate or poor); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.63 to 1.40] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by IMDC risk group (favorable vs. intermediate or poor)

3. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated a confirmed complete response (CR: Disappearance of all target lesions) or confirmed partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR as assessed by blinded independent central review was presented.
Time Frame: Up to approximately 27 months
Population: The analysis population consisted of all randomized participants based on the treatment group to which they were randomized who experienced a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 18 | 18
Months | 16.1 [6.5 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [3.8 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

4. Secondary Outcome: Clinical Benefit Rate (CBR) Per RECIST 1.1 as Assessed by BICR
Description: CBR is defined as the percentage of participants who have a complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) or stable disease (SD: Neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.) ≥6 months per RECIST 1.1. The percentage of participants with CBR will be presented.
Time Frame: Up to approximately 27 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Percentage of Participants | 41.0 [30.0 to 52.7] | 47.4 [35.8 to 59.2]
Statistical Analysis 1: Comparison: Belzutifan 200 mg vs Belzutifan 120 mg; Test type: Other — One-sided nominal p-value, difference in percentage and associated 95% CIs were based on Miettinen & Nurminen method stratified by IMDC risk group (favorable vs. intermediate or poor); p = 0.7832, Miettinen & Nurminen method; Miettinen & Nurminen method = -6.3, 95% CI 2-sided [-21.7 to 9.4]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 27 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Months | NA [20.6 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [22.0 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Belzutifan 200 mg vs Belzutifan 120 mg; Test type: Other; p = 0.6448, Log Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; One-sided nominal p-value based on log-rank test stratified by IMDC risk group (favorable vs. intermediate or poor); Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.65 to 1.90] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one or more AEs was presented.
Time Frame: Up to approximately 27 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Number of Participants | 77 | 75

7. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE was presented.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 78 | 76
Number of Participants | 11 | 4

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Belzutifan
Description: Blood samples were obtained at designated time points for the determination of the Cmax of belzutifan.
Time Frame: Weeks 1 and 3 on Day 1: predose and 1, 2, and 4 hours. Week 5 on Day 1: predose only
Population: The analysis population consisted of all randomized participants based on the treatment group to which they were randomized who had at least 1 measurable belzutifan concentration observation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 77 | 75
ng/mL | 2512 (86) | 1518 (97)

9. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Belzutifan
Description: Blood samples were obtained at designated time points for the determination of the Ctrough of belzutifan.
Time Frame: Weeks 1 and 3 on Day 1: predose and 1, 2, and 4 hours. Week 5 on Day 1: predose only
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
Number analyzed (Participants) | 77 | 75
ng/mL | 513 (158) | 296 (159)

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Belzutifan 200 mg | Belzutifan 120 mg
All-Cause Mortality (participants affected / at risk) | 28/78 | 25/76
Serious Adverse Events (participants affected / at risk) | 33/78 | 33/76
Other Adverse Events (participants affected / at risk) | 75/78 | 74/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belzutifan 200 mg (N=78) | Belzutifan 120 mg (N=76)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belzutifan 200 mg (N=78) | Belzutifan 120 mg (N=76)
Anaemia (Blood and lymphatic system disorders) | 64 (71) | 58 (77)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Vision blurred (Eye disorders) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 9 (12)
Constipation (Gastrointestinal disorders) | 8 (10) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 7 (13) | 10 (14)
Nausea (Gastrointestinal disorders) | 18 (26) | 27 (34)
Vomiting (Gastrointestinal disorders) | 7 (15) | 9 (12)
Asthenia (General disorders) | 8 (10) | 1 (1)
Chest pain (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 42 (48) | 40 (47)
Oedema peripheral (General disorders) | 18 (26) | 18 (21)
Pyrexia (General disorders) | 7 (8) | 7 (10)
COVID-19 (Infections and infestations) | 9 (9) | 11 (11)
Urinary tract infection (Infections and infestations) | 3 (5) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 8 (9)
Alanine aminotransferase increased (Investigations) | 10 (11) | 11 (19)
Aspartate aminotransferase increased (Investigations) | 10 (15) | 11 (18)
Blood creatinine increased (Investigations) | 10 (13) | 12 (14)
Blood glucose increased (Investigations) | 4 (4) | 3 (7)
Blood sodium decreased (Investigations) | 4 (6) | 2 (3)
Haemoglobin decreased (Investigations) | 8 (10) | 5 (6)
Lymphocyte count decreased (Investigations) | 4 (6) | 5 (8)
Weight decreased (Investigations) | 4 (5) | 4 (4)
Weight increased (Investigations) | 6 (6) | 6 (8)
Decreased appetite (Metabolism and nutrition disorders) | 12 (16) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (5) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 18 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 14 (18)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (10)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 11 (13) | 15 (19)
Headache (Nervous system disorders) | 17 (23) | 22 (25)
Haematuria (Renal and urinary disorders) | 5 (10) | 6 (8)
Proteinuria (Renal and urinary disorders) | 1 (1) | 7 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 18 (21)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 17 (24)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Hypertension (Vascular disorders) | 11 (16) | 8 (10)
Hypotension (Vascular disorders) | 2 (2) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT04489771/Prot_SAP_000.pdf